CLINICAL TRIAL: NCT01711710
Title: Clinical Trial to Evaluate the Safety and Efficacy of Cohesive Silicone Gel-Filled Breast Implant (CoSBI) in Women Aged 22 and Over With Breast Reconstruction or Augmentation Mammoplasty.
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of Breast Implant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: HansBiomed Co.,Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-2010-095; E-1005-049-001 (Other: IRB)
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer; reconstruction; augmentation; cohesive silicone gel; breast implant; rupture; capsular contracture
MeSH Terms: conditions — Breast Neoplasms; Rupture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cohesive Gel Breast Implant (Experimental): Cohesive Silicone Gel-Filled Breast Implant
  Interventions: Device: Cohesive Gel Breast Implant

INTERVENTIONS:
Device: Cohesive Gel Breast Implant — Cohesive Silicone Gel-Filled Breast Implant insert under the submuscular with axillary incision in breast augmentation mammoplasty.
  Remove tissue expander and insert Cohesive Silicone Gel-Filled Breast Implant in breast reconstruction.
  Other Names: Cohesive Silicone Gel-Filled Breast Implant(CoSBI)

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of Cohesive Silicone Gel-Filled Breast Implant (CoSBI) produced by HansBiomed co.,Ltd. in breast reconstruction or augmentation

ELIGIBILITY:
Inclusion Criteria:

* Over 22 years of age
* Subjects who want breast augmentation reconstruction following breast cancer, congenital or accidental unbalanced breast size
* Negative pregnancy test in fertile women
* Subjects who voluntarily decided the participation of the study and signed the informed consent
* Subjects who can understand and comply with the instructions and participate during the entire period of the trial

Exclusion Criteria:

* previous breast reconstruction or augmentation history
* self -immune disease
* uncontrolled active infectious disease
* unable to insert beast implant due to radiotherapy
* Patients who have recurrent breast cancer or do not treat effectively their cancer
* Keloid
* Abnormal blood test or ECG result for general anesthesia
* Patients who cannot MRI scan due to having Metallic substance in the body or Claustrophobia
* Aesthetic addiction, drug abuse, alcohol abuse
* Patients who are not eligible for this study at the medical discretion of the Principal Investigator or Sub-investigator

Min Age: 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2010-10-30; Primary Completion 2014-10-30 (Actual); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
a rate of rupture of 1% | 2 years
  All the subjects have been monitored for 2 years and will be checked MRI to define rupture at 6month, 1 year and 2year after the breast implant.
a rate of capsular contracture of 5% | 2 years
  The Baker classification that divided into 4 stages will be used as a reference to evaluate the capsular contracture. Only stage 3 and 4 will be confirmed as capsular contracture.

SECONDARY OUTCOMES:
a rate of connective tissue disease | 2 years
  Connective tissue disease include hair loss, erythema, photosensitivity, dry eye syndrome,myalgia,neuralgia,arthralgia, etc.
Changes in bust girth and actual measured bra-cup size | 2 years
  Bra cup size can be determined by measuring right or left bust circumference over the nipple.
  6 inch= doubleA, 7inch=A, 8inch= B, 9inch=C, 10inch=D, 11inch=E Bust girth means bust circumference line . It can be determined by measuring around the women's torso over the fullest part of the breasts.
Change in life satisfaction | 2 years
  The subject questionaire including Rosenberg Self Esteem Scale,Body Esteem Scale,Survey of Functional-36 Status Survey will be assessed at 6month, 1year and 2year after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Chanyeong Heo, Ph. D, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Samsung Medical Center, Seoul